CLINICAL TRIAL: NCT07366528
Title: Adjuvant Oxaliplatin Plus S-1 Versus Docetaxel Plus S-1 for Stage III Gastric Cancer After D2 Gastrectomy (DRAGON-Adjuvant): a Multicenter, Open-label, Phase 3, Randomized, Non-inferiority Study
Brief Title: Adjuvant Oxaliplatin Plus S-1 Versus Docetaxel Plus S-1 for Stage III Gastric Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Clinical Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRAGON-Adjuvant/2025-No.675
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Gastric Cancer (GC); Adjuvant Chemotherapy; Stage 3 Cancer; Docetaxel; Oxaliplatin
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — Oxaliplatin; S 1 (combination); Docetaxel

STUDY DESIGN:
Intervention Model Description: SOX group: eight 3-week cycles of intravenous oxaliplatin (130mg/m2 on day 1 for each cycle) with orally S-1 dose dependent on body surface area (<1.24 m2, 40mg twice a day; 1.25-1.5 m2, 50mg twice a day; >1.5m2 60mg twice a day, days 1 to 14 of each cycle).
  DS group: S-1 on days 1 to 14 of a 3-week cycle during the first cycle. During the second to seventh cycles, patients received intravenous infusion of docetaxel (40mg/m2) on day 1 of each cycle and S-1 on days 1 to 14 of a 3-week cycle. After the eighth cycle, treatment with S-1 continued on days 1 to 28 of 6-week cycles for up to 1 year.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxaliplatin plus S-1 (Experimental): Patients will be treated with oxaliplatin plus S-1 as adjuvant therapy
  Interventions: Drug: Oxaliplatin plus S-1
- Docetaxel plus S-1 (Active Comparator): Patients will be treated with docetaxel plus S-1 as adjuvant therapy
  Interventions: Drug: Docetaxel plus S-1

INTERVENTIONS:
Drug: Oxaliplatin plus S-1 — SOX group: eight 3-week cycles of intravenous oxaliplatin (130mg/m2 on day 1 for each cycle) with orally S-1 dose dependent on body surface area (<1.24 m2, 40mg twice a day; 1.25-1.5 m2, 50mg twice a day; >1.5m2 60mg twice a day, days 1 to 14 of each cycle).
  Arms: Oxaliplatin plus S-1
Drug: Docetaxel plus S-1 — DS group: S-1 on days 1 to 14 of a 3-week cycle during the first cycle. During the second to seventh cycles, patients received intravenous infusion of docetaxel (40mg/m2) on day 1 of each cycle and S-1 on days 1 to 14 of a 3-week cycle. After the eighth cycle, treatment with S-1 continued on days 1 to 28 of 6-week cycles for up to 1 year.
  Arms: Docetaxel plus S-1

SUMMARY:
This is a multicenter, open-label, phase 3, randomized, non-inferiority study aimed to investigate the effect on disease-free survival of adjuvant chemotherapy with oxaliplatin plus S-1 compared with adjuvant chemotherapy with docetaxel plus S-1 after D2 gastrectomy in patients with stage III gastric cancer.

DETAILED DESCRIPTION:
In gastric cancer, adjuvant chemotherapy that can reduce the risk of recurrence and improve patient survival has been a standard of care for gastric cancer patients with pathological stage II-III after D2 gastrectomy and R0 resection. Currently, oxaliplatin plus S-1 (SOX) or docetaxel plus S-1 (DS) have been recommended as adjuvant therapy for stage III gastric cancer patients, based on the results of RESOLVE trial and JACCRO GC-07 trial, respectively. However, due to the different study design and patient enrollment, the efficacy of these two regimens can hardly be compared directly. The safety profiles and treatment period of the two regimens can be factors to guide regimen selection. For SOX regimen, oxaliplatin-related peripheral neuropathy and allergy are clinical concerned issues. Although frequency of similar toxicities of docetaxel is lower, S-1 should be administrated for 12 months after surgery in the DS regimen. Prolonged treatment period also increases the risk of treatment-related toxicities and impairs patients' adherence. There is necessary to compare these two regimens directly. In this study, gastric cancer patients who undergo D2 gastrectomy and achieve R0 resection with pathological stage III (IIIA, IIIB, IIIC) will be randomized and treated with SOX or DS regimen. In SOX group, eight 3-week cycles of intravenous oxaliplatin (130mg/m2 on day 1 for each cycle) with orally S-1 dose dependent on body surface area (<1.24 m2, 40mg twice a day; 1.25-1.5 m2, 50mg twice a day; >1.5m2 60mg twice a day, days 1 to 14 of each cycle). In DS group, S-1 dose is also determined by body surface area. Patients are treated with S-1 on days 1 to 14 of a 3-week cycle during the first cycle. During the second to seventh cycles, patients received intravenous infusion of docetaxel (40mg/m2) on day 1 of each cycle and S-1 on days 1 to 14 of a 3-week cycle. After the eighth cycle, treatment with S-1 continued on days 1 to 28 of 6-week cycles for up to 1 year. Patients will be followed up for 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 80 years old, male and female
2. histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction
3. patients underwent standard D2 gastrectomy and achieved R0 resection, and had no systemic therapy like neoadjuvant therapy
4. American Joint Committee on Cancer stage IIIA (T2N3a, T3N2, T4aN1, T4aN2, T4bN0), IIIB (T1N3b, T2N3b, T3N3a, T4aN3a, T4bN1, T4bN2), IIIC (T3N3b, T4aN3b, T4bN3a, T4bN3b), and has Lauren classification
5. with no evidence of metastatic disease
6. ECOG 0 to 1
7. Enough organ functions that can tolerate treatment: Absolute neutrophil count (ANC) ≥1.5x109/L, White blood count ≥3.5x109/L, Platelets ≥75x109/L, Hemoglobin (Hb) ≥80g/L, ALT/AST ≤2.5x ULN (for patient with liver metastasis ALT/AST ≤5x ULN), Serum bilirubin ≤1.5x ULN, Serum creatinine ≤1.5x ULN.
8. Woman of childbearing age should contracept for at least one month before screening and commit to using contraception throughout the entire study period and for the specified time after the study ends.
9. Signed informed consent and willing to follow the study protocol

Exclusion Criteria:

1. other primary malignancies, except for cured skin tumors or cervical carcinoma in situ
2. severe complications that may lead to an expected survival time less than 5 years
3. uncontrollable comorbidities, such as infectious disease, chronic diseases like hypertension, diabetes, heart diseases.
4. allergic to study medication
5. bowel obstruction or other conditions affecting oral administration
6. organ functions that cannot tolerate study treatment
7. other conditions that patients are unsuitable for this study assessed by the investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | From randomization to 3 years after randomization
  Defined as the proportion of patients who remain free from recurrence of the original gastric cancer, development of a new gastric cancer, or death from any cause at 3 years after randomization.

SECONDARY OUTCOMES:
5-year overall survival rate | From randomization to 5 years after randomization
  Defined as the proportion of patients who remain survival at 5 years after randomization.
Safety profiles | through treatment completion, an average of 6 months
  Adverse events during treatment
Recurrence sites | From randomization to 3 years after randomization
  Organs involved in tumor metastasis and recurrence

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Yuebei People's Hospital, Shaoguan, Guandong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Renji Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided